CLINICAL TRIAL: NCT06830213
Title: Investigation of the Validity, Reliability and Responsiveness of the BETY-Biopsychosocial Questionnaire in Familial Mediterranean Fever
Brief Title: Investigation of the Validity, Reliability and Responsiveness of the BETY-BQ in FMF
Status: Not yet recruiting | Type: Observational
Sponsor: Aysima Barlak (Other)
Responsible Party: Sponsor-Investigator, Aysima Barlak, PT, Hacettepe University
Organization: Hacettepe University (Other)
Other Study IDs: SBA 24/1114
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-12

CONDITIONS: Familial Mediterranean Fever (FMF )
Keywords: Familial Mediterranean Fever; biopsychosocial; depression; social isolation; pain; sleep; functionality
MeSH Terms: conditions — Familial Mediterranean Fever; Depression; Social Isolation; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Questionnaire study — Questionnaire application

SUMMARY:
FMF is associated with many different clinical entities. The disease appears to be associated with many diseases and/or syndromes with common features of genetic predisposition, immune dysfunction and autoinflammation. Pericardial inflammation, cardiovascular conditions such as ischaemic heart disease, other rheumatic diseases such as ankylosing spondylitis (AS), vasculitis, especially Behçet's disease, malignancy and infertility are often associated with FMF. Early detection of these associations makes it possible to improve the management and prognosis of patients with FMF.

The chronic nature of the disease, as in other chronic diseases, includes problems such as pain, fatigue, sleep problems, loss of function, anxiety, depression and social isolation. This complex structure is accompanied by a picture in which inflammatory processes are triggered.

When the literature is examined, it is emphasised that chronic diseases with multifaceted symptoms require evaluation and methods that include all these biopsychosocial features. On the other hand, although it is stated that the common goal of non-pharmacological treatments is to contribute to biopsychosocial improvement in the patient, it is emphasised that evaluations with biopsychosocial content are insufficient. This situation causes the need for scales that provide an assessment from a holistic perspective in chronic diseases.

Cognitive Exercise Therapy Approach (BETY) is an innovative exercise approach developed on the basis of biopsychosocial model on individuals with rheumatism. The parameters that constitute the innovation are detailed under four headings: function-oriented core stabilisation exercises, information management in pain, information management in mood, and information management in sexuality. This method has a unique scale that offers biopsychosocial assessment. The Cognitive Exercise Therapy Approach - Biopsychosocial Questionnaire (BETY-BQ) was created by receiving feedback from individuals with rheumatism who participated in BETY exercise training 3 days a week for many years, expressing the improvement characteristics they experienced by participating in exercise sessions. The BETY-BQ evaluates the individual biopsychosocially with six sub-headings: pain, functionality-fatigue, emotion-state, sociability, sexuality and sleep.

The validity, reliability and sensitivity of the BETY-BQ have been demonstrated in many rheumatic diseases such as rheumatoid arthritis, fibromyalgia, psoriatic arthritis, systemic lupus erythematosus, ankylosing spondylitis, knee osteoarthritis, primary Sjögren's syndrome. Currently, it is clear that there is a need for scales that offer biopsychosocial assessment for individuals diagnosed with rheumatism, where biopsychosocial approaches are recommended in EULAR recommendations. BETY-BQ is included in the EULAR library as a biopsychosocial status measurement tool. This study will investigate the validity, reliability and responsiveness of the BETY-BQ, a biopsychosocial assessment tool, in individuals diagnosed with Familial Mediterranean Fever.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of Familial Mediterranean Fever
* Being literate
* Being 18 years of age or older
* Having read and signed the informed consent

Exclusion Criteria:

* History of major psychiatric illness
* Malignant disease
* History of peripheral vascular disease or neuropathy
* Not volunteering for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals who come to the university hospital for routine controls.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-18 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
BETY-Biopsychosocial Questionnaire | 3 mounths
  The biopsychosocial status of the individual is assessed with questions about pain, functionality, mood, sociability, sexuality, and sleep status. Each question consists of 30 items scored between 0-120 as '0 (never), 1 (yes rarely), 2 (yes sometimes), 3 (yes often), 4 (yes always)'. A high score indicates poor biopsychosocial status

SECONDARY OUTCOMES:
Hospital Anxiety Depression Scale | 3 mounths
  It consists of 14 items, 7 of which assess anxiety, and the other 7 determine depression. Each item is scored between 0-3, and the total is scored between 0-21. High scores indicate poor anxiety and depression levels.
Health Assessment Questionnaire | 3 mounths
  The Health Assessment Questionnaire evaluates the functionality of the individual using eight parameters and 20 items. The parameters are classified as dressing, standing, eating, walking, hygiene, reaching, grasping, and other activities. Each item is scored as 0 (without any difficulty), 1 (with some difficulty), 2 (with a lot of difficulty), and 3 (unable to do at all). The total score is between 0-3, with a high score indicating low functionality.
Short Form - 36 | 3 mounths
  The SF-36 is a patient-orientated assessment scale created in the United States of America that allows for general health screening. Each sub-parameter is scored between 0 and 100 points and a high score indicates good health status. The SF-36 scale has 8 sub-parameters including general health perception, physical function, social function, pain, mental health, role difficulties due to physical causes, role difficulties due to emotional causes and vitality and includes 11 questions with a total of 36 items.
Pain Catastrophizing Scale | 3 mounths
  This scale, developed by Sullivan et al. serves to measure the extent to which individuals catastrophise pain and the exaggerated negative mental reaction they show to current or anticipated painful experience. The scale consists of 13 items. Each item is scored as never=0, slightly=1, moderately=2, greatly=3 and always=4. A high total score indicates a high degree of catastrophising of pain.
Fatigue Severity Scale | 3 mounths
  It is a scale that evaluates fatigue and consists of 9 questions. Each item is scored between 0 and 7. The total score is divided by 9, and if the average is <4, no fatigue is assessed, and if ≥4, fatigue is assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No